CLINICAL TRIAL: NCT01194414
Title: A Randomized, Double-blind, Parallel Group Study of the Safety and Effect on Clinical Outcome of Tocilizumab SC Versus Tocilizumab IV, in Combination With Traditional Disease Modifying Anti-rheumatic Drugs (DMARDs), in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Compare Subcutaneous Versus Intravenous Administration of RoActemra/Actemra (Tocilizumab) in Participants With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA22762; 2010-018375-22
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2013-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Tocilizumab SC (Experimental): Participants received tocilizumab 162 mg subcutaneous (SC) injection weekly plus placebo to tocilizumab intravenous (IV) infusion every 4 weeks for a total of 24 weeks in the double-blind period. Participants continued to receive tocilizumab 162 mg SC injection weekly for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose continued throughout the study.
  Interventions: Drug: tocilizumab SC; Drug: placebo to tocilizumab IV; Drug: Disease-modifying antirheumatic drugs (DMARDs)
- Tocilizumab IV (Experimental): Participants received tocilizumab 8 mg/kg infusion (IV) every 4 weeks plus placebo to tocilizumab SC injection weekly for a total of 24 weeks in the double-blind period. Participants continued to receive tocilizumab 8 mg/kg IV infusion every 4 weeks for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose continued throughout the study.
  Interventions: Drug: tocilizumab IV; Drug: placebo to tocilizumab SC; Drug: Disease-modifying antirheumatic drugs (DMARDs)
- Tocilizumab SC Then Tocilizumab IV (Experimental): Participants who received tocilizumab 162 mg subcutaneous (SC) injection weekly plus placebo to tocilizumab IV infusion every 4 weeks for 24 weeks in double blind treatment period switched to tocilizumab 8 mg/kg IV infusion every 4 weeks for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose continued throughout the study.
  Interventions: Drug: tocilizumab SC; Drug: tocilizumab IV; Drug: placebo to tocilizumab IV; Drug: Disease-modifying antirheumatic drugs (DMARDs)
- Tocilizumab IV Then Tocilizumab SC (Experimental): Participants who received tocilizumab 8 mg/kg infusion (IV) every 4 weeks plus placebo to tocilizumab SC injection weekly in double blind treatment period switched to tocilizumab 162 mg SC injection weekly for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose will be continued throughout the study.
  Interventions: Drug: tocilizumab SC; Drug: tocilizumab IV; Drug: placebo to tocilizumab SC; Drug: Disease-modifying antirheumatic drugs (DMARDs)

INTERVENTIONS:
Drug: tocilizumab SC — Tocilizumab supplied in a single-use pre-filled syringe, with a needle safety device, delivering 162 mg/0.9 mL solution for subcutaneous injection once a week.
  Other Names: RoActemra/Actemra
  Arms: Tocilizumab IV Then Tocilizumab SC; Tocilizumab SC; Tocilizumab SC Then Tocilizumab IV
Drug: tocilizumab IV — Tocilizumab supplied in vials as a sterile solution for 8 mg/kg intravenous infusion every 4 weeks.
  Other Names: RoActemra/Actemra
  Arms: Tocilizumab IV; Tocilizumab IV Then Tocilizumab SC; Tocilizumab SC Then Tocilizumab IV
Drug: placebo to tocilizumab SC — Placebo tocilizumab supplied as a single-use pre-filled syringe with a needle safety device, delivering 0.9 mL sodium chloride for subcutaneous injection once a week for 24 weeks in the double-blind period.
  Arms: Tocilizumab IV; Tocilizumab IV Then Tocilizumab SC
Drug: placebo to tocilizumab IV — Placebo to tocilizumab supplied as a solution in 10 mL vials containing polysorbate 80 and sucrose in water for infusion every 4 weeks for a total of 24 weeks in the double-blind period.
  Arms: Tocilizumab SC; Tocilizumab SC Then Tocilizumab IV
Drug: Disease-modifying antirheumatic drugs (DMARDs) — stable dose as prescribed

SUMMARY:
This randomized, double-blind, parallel group study compares the efficacy and safety of subcutaneous (sc) versus intravenous (iv) administration of tocilizumab in participants with moderate to severe active rheumatoid arthritis. Participants were randomized to receive either tocilizumab 162 mg sc weekly plus iv placebo every 4 weeks, or tocilizumab 8 mg/kg iv every 4 weeks plus sc placebo weekly during the double-blind period from baseline to Week 24. The double-blind period was followed by a 72-week open-label treatment with some switching of sc and iv administration. No placebo was administered in the open-label phase. Participants continued on their stable dose of disease-modifying antirheumatic drugs (DMARDs) throughout the study. Anticipated time on study treatment was 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, ≥ 18 years of age
* Rheumatoid arthritis of ≥ 6 months duration, according to American College of Rheumatology (ACR) criteria
* Swollen joint count (SJC) ≥ 4 (66 joint count), tender joint count (TJC) ≥ 4 (68 joint count) at screening and baseline
* Inadequate response to current DMARD therapy
* Permitted DMARDs must be at stable dose for ≥ 8 weeks prior to baseline
* Oral corticosteroids (≤ 10 mg/day prednisone or equivalent) and NSAIDs (up to maximum recommended dose) must be at stable dose for ≥ 4 weeks prior to baseline

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Rheumatic autoimmune disease other than RA
* Functional class IV (ACR classification)
* Diagnosis of juvenile idiopathic arthritis (JIA) or juvenile rheumatoid arthritis (JRA) and/or RA before the age of 16
* Prior history of or current inflammatory joint disease other than RA
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* Previous treatment with tocilizumab
* Active current or history of recurrent infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1262 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (190):
- United States (51):
  - Huntsville, Alabama
  - Tuscaloosa, Alabama
  - Tucson, Arizona
  - Long Beach, California
  - Los Angeles, California
  - Upland, California
  - Van Nuys, California
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Delray Beach, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Pinellas Park, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Morton Grove, Illinois
  - Wichita, Kansas
  - Monroe, Louisiana
  - Petoskey, Michigan
  - Saint Claire Shores, Michigan
  - Eagan, Minnesota
  - Florissant, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Clifton, New Jersey
  - Manalapan, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Orchard Park, New York
  - Asheville, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Olympia, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Wenatchee, Washington
- Argentina (2):
  - Buenos Aires
  - Rosario
- Australia (7):
  - Adelaide
  - Clayton
  - Geelong
  - Hobart
  - Malvern East
  - Maroochydore
  - New Lambton
- Brazil (5):
  - Curitiba
  - Goiânia
  - Juiz de Fora
  - Porto Alegre
  - São Paulo
- Sofia, Bulgaria
- Canada (15):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Ottawa, Ontario
  - St. Catharines, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Rimouski, Quebec
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
- Colombia (2):
  - Barranquilla
  - Bogotá
- France (8):
  - Bordeaux
  - Le Mans
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Strasbourg
  - Toulouse
- Germany (15):
  - Bad Bramstedt
  - Berlin
  - Cologne
  - Dresden
  - Essen
  - Freiburg im Breisgau
  - Gommern
  - Heidelberg
  - Herne
  - Hildesheim
  - Ludwigshafen
  - Osnabrück
  - Ratingen
  - Rostock
  - Würzburg
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Italy (12):
  - Arenzano
  - Bergamo
  - Catania
  - Cona (ferrara)
  - Genova
  - Napoli
  - Pavia
  - Pisa
  - Potenza
  - Reggio Emilia
  - Udine
  - Varese
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Mexico (11):
  - Culiacán
  - Guadalajara
  - León
  - Mexico Ctiy
  - Mérida
  - Miexico City
  - Morelia
  - Obregón
  - Querétaro
  - Saltillo
  - Torreón
- New Zealand (4):
  - Auckland
  - Hamilton
  - Tauranga
  - Wellington
- Lima, Peru
- Philippines (3):
  - Cebu
  - Manila
  - Quezon
- Poland (4):
  - Bialystok
  - Lublin
  - Poznan
  - Warsaw
- Ponce, Puerto Rico
- Romania (2):
  - Bucharest
  - Iași
- Russia (6):
  - Moscow
  - Novosibirsk
  - Ryazan
  - Saint Petersburg
  - Ulyanovsk
  - Yaroslavl
- Singapore, Singapore
- South Africa (5):
  - Cape Town
  - Durban
  - Parktown
  - Port Elizabeth
  - Stellenbosch
- Spain (12):
  - A Coruña
  - Barakaldo
  - Bilbao
  - Madrid
  - Málaga
  - Mérida
  - San Cristóbal de La Laguna
  - Santander
  - Santiago de Compostela
  - Seville
  - Torrelavega
  - Valencia
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- United Kingdom (14):
  - Cambridge
  - Cannock
  - Coventry
  - Eastbourne
  - Exeter
  - Harrogate
  - Ipswich
  - London
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - Newcastle upon Tyne
  - Northampton
  - Nottingham
  - Westcliffe-on-sea

REFERENCES:
- [Derived] Burmester GR, Rubbert-Roth A, Cantagrel A, Hall S, Leszczynski P, Feldman D, Rangaraj MJ, Roane G, Ludivico C, Bao M, Rowell L, Davies C, Mysler EF. Efficacy and safety of subcutaneous tocilizumab versus intravenous tocilizumab in combination with traditional DMARDs in patients with RA at week 97 (SUMMACTA). Ann Rheum Dis. 2016 Jan;75(1):68-74. doi: 10.1136/annrheumdis-2015-207281. Epub 2015 Jun 8. PMID 26056119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1262 participants at 209 centers in 25 countries were randomized into the study.
Groups:
- Tocilizumab IV Then Tocilizumab SC: Participants who received tocilizumab 8 mg/kg infusion (IV) every 4 weeks plus placebo to tocilizumab SC injection once a week in double blind treatment period switched to tocilizumab 162 mg SC injection weekly for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose will be continued throughout the study.
Period: 24 Weeks Double Blind Period
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Started | 631 | 631 | 0 | 0
Per Protocol Population | 558 | 537 | 0 | 0
Completed | 572 | 564 | 0 | 0
Not Completed | 59 | 67 | 0 | 0
Not completed — Insufficient Therapeutic Response | 11 | 8 | 0 | 0
Not completed — Subject/legal Guardian Decision | 9 | 5 | 0 | 0
Not completed — Protocol Violation | 5 | 3 | 0 | 0
Not completed — Physician Decision to Withdraw Subject | 0 | 5 | 0 | 0
Not completed — Pregnancy | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Adverse Event | 28 | 40 | 0 | 0
Not completed — Anaphylaxis or Hypersensitivity Reaction | 2 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: 72 Weeks Open Label Extension
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Started | 524 | 377 | 48 | 186
Completed | 445 | 311 | 40 | 160
Not Completed | 79 | 66 | 8 | 26
Not completed — Randomized but not Treated | 3 | 5 | 0 | 0
Not completed — Subject/legal Guardian Decision | 20 | 14 | 1 | 6
Not completed — Insufficient Therapeutic Response | 9 | 11 | 2 | 3
Not completed — Lost to Follow-up | 4 | 3 | 2 | 1
Not completed — Physician Decision to Withdraw Subject | 3 | 5 | 0 | 0
Not completed — Pregnancy | 1 | 3 | 1 | 1
Not completed — Other | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 35 | 21 | 2 | 12
Not completed — Anaphylaxis or Hypersensitivity Reaction | 1 | 1 | 0 | 0
Not completed — Death | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab SC: Participants received tocilizumab 162 mg subcutaneous (SC) injection weekly plus placebo to tocilizumab intravenous (IV) infusion every 4 weeks for a total of 24 weeks in the double-blind period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose beginning at least 8 weeks prior to baseline were a requirement of the study.
- Tocilizumab IV: Participants received tocilizumab 8 mg/kg infusion (IV) every 4 weeks plus placebo to tocilizumab SC injection weekly for a total of 24 weeks in the double-blind period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose beginning at least 8 weeks prior to baseline were a requirement of the study.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab SC | Tocilizumab IV | Total
Number analyzed (Participants) | 631 | 631 | 1262
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.35) [18 to 83] | 52.8 (12.53) [18 to 86] | 52.7 (12.44) [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 520 | 521 | 1041
  Male | 111 | 110 | 221

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology Criteria (ACR20) Response at Week 24
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the five additional ACR core set variables: Patient's Assessment of Pain over the previous 24 hours using a Visual Analog Scale (VAS) where left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and acute-phase reactant (either C-reactive protein [CRP] or Erythrocyte Sedimentation Rate [ESR]).
Time Frame: Baseline, 24 weeks
Population: Per Protocol Population included all randomized participants who received study drug and had no major protocol violations. Last Observation Carried Forward was used for missing joint counts, no imputation for other ACR components. CRP will be used primarily for calculation of the ACR response. If missing, the ESR will be used for that participant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 558 | 537
Percentage of participants | 69.4 [65.5 to 73.2] | 73.4 [69.6 to 77.1]

2. Primary Outcome: Percentage of Participants With Adverse Events, Serious Adverse Events and Clinically Significant Laboratory Assessments
Time Frame: Baseline to up to 3 months after last dose of study drug (approximately up to 2 years)
Population: The safety population includes all participants who received at least one dose of study drug, whether re-randomized or not, and who had at least one post-dose safety assessment. Data are included from double blind and open label (OL) periods in the SC and IV arms but only from the OL period in IV-SC and SC-IV switch arms.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 631 | 631 | 48 | 186
percentage of participants
  Adverse Events (AEs) | 91.6 | 87.8 | 81.3 | 86.6
  Serious Adverse Events (SAEs) | 13.9 | 12.7 | 12.5 | 11.3
  Clinically Significant Laboratory Assessments | 37.7 | 28.2 | 25.0 | 19.4

3. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology Criteria (ACR50) Response at Week 24
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the five additional ACR core set variables: Patient's Assessment of Pain over the previous 24 hours using a Visual Analog Scale (VAS) where left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and acute-phase reactant (either C-reactive protein or Erythrocyte Sedimentation Rate).
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 558 | 537
Percentage of participants | 47.0 | 48.6

4. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology Criteria (ACR70) Response at Week 24
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the five additional ACR core set variables: Patient's Assessment of Pain over the previous 24 hours using a Visual Analog Scale (VAS) where left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and acute-phase reactant (either C-reactive protein or Erythrocyte Sedimentation Rate).
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 558 | 537
Percentage of participants | 24.0 | 27.9

5. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 (DAS28) Remission at Week 24
Description: The DAS28 (ESR) score is a measure of the subject's disease activity. It is calculated using the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity VAS where left side of the line 0=no disease activity to right side of the line 100=extreme disease activity and ESR. DAS28-(ESR) total scores range from 0 - 10. Remission is defined as achieving a DAS28-ESR score of less than 2.6.
Time Frame: Week 24
Population: Participants from the Per Protocol Population (randomized participants who received study drug and had no major protocol violations) with data available for analysis. Missing SJC and TJC will be imputed using the last post-baseline value for the patient (LOCF). No imputation for missing ESR or patient's global assessment of disease activity.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 516 | 498
Percentage of participants | 38.4 | 36.9

6. Secondary Outcome: Percentage of Participants Achieving a Decrease of ≥ 0.3 in the Health Assessment Questionnaire-Disability Index (HAQ-DI) From Baseline to Week 24
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a participant completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. A decrease indicates improvement.
Time Frame: Baseline, 24 Weeks
Population: Participants from the Per Protocol Population (all randomized participants who received study drug and had no major protocol violations) with data available for analysis. No imputation of missing scores will be made other than for missing baseline scores, for which last score prior to defined protocol baseline time window will be carried forward.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 515 | 500
Percentage of participants | 65.2 | 67.4

7. Secondary Outcome: Percentage of Participants Who Withdrew Because of Lack of Therapeutic Response at Week 24
Description: The percentage of participants who withdrew from the study because they were not responding to treatment with the study drug.
Time Frame: 24 Weeks
Population: Per Protocol Population included all randomized participants who received study drug and had no major protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 558 | 537
Percentage of participants | 1.8 | 0.9

8. Secondary Outcome: Percentage of Participants With American College of Rheumatology Criteria (ACR20, ACR50, ACR70) at Week 97
Description: ACR20, ACR50 and ACR70: ≥20%, ≥50% and ≥70% reduction from baseline for both TJC68 and SJC66, as well as for 3 of 5 additional ACR variables: Patient's Assessment of Pain in last 24 hours using a Visual Analog Scale (VAS) (0=no pain and 100=unbearable pain); Patient's and Physician's Global Assessment of Disease Activity in last 24 hours using a VAS (0=no disease activity and100=maximum disease activity); Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and acute-phase reactant (either CRP or ESR). CRP was used for calculation of ACR. If missing, ESR was used. LOCF was used for missing joint counts, no imputation for other ACR components.
Time Frame: Week 97
Population: Re-Randomized Intent-to-Treat Population (ITT Population) included all participants who completed double blind period and were re-randomized at Week 24, received at least 1 dose of study drug. Here, number of participants analyzed is the participants for whom parameter was collected.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 451 | 317 | 40 | 165
percentage of participants
  ACR20 | 83.6 | 83.3 | 82.5 | 88.5
  ACR50 | 65.4 | 62.5 | 57.5 | 67.3
  ACR70 | 44.8 | 42.0 | 37.5 | 47.3

9. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 (DAS28) Remission at Week 97
Description: The DAS28 (ESR) score is a measure of the subject's disease activity. It is calculated using the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity VAS where left side of the line 0=no disease activity to right side of the line 100=extreme disease activity and ESR. DAS28-(ESR) total scores range from 0 - 10. Remission is defined as achieving a DAS28-ESR score of less than 2.6. LOCF used for tender and swollen joint counts, no imputation used for ESR and Patient's Global Assessment of Disease Activity VAS.
Time Frame: Week 97
Population: ITT Population included all participants who completed double blind period and were re-randomized at Week 24 and received at least one dose of study drug. If ESR=0 then ESR=1 is substituted into the DAS28 calculation to enable a non-missing DAS28 score. Here, number of participants analyzed is the participants for whom parameter was collected.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 446 | 306 | 40 | 162
percentage of participants | 53.4 | 46.4 | 50.0 | 55.6

10. Secondary Outcome: Percentage of Participants Achieving a Decrease of ≥0.3 in the Health Assessment Questionnaire-Disability Index (HAQ-DI) From Baseline to Week 97
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. A decrease indicates improvement. No imputation of missing scores was made other than for missing baseline scores, for which last score prior to baseline will be carried forward. For participants who prematurely withdrew, data collected at withdrawal visit was used and data thereafter is missing.
Time Frame: Baseline, Week 97
Population: ITT Population included all participants who completed double blind period and were re-randomized at Week 24 and received at least one dose of study drug. Here, number of participants analyzed is the participants for whom parameter was collected.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 445 | 317 | 39 | 162
percentage of participants | 72.4 | 69.1 | 56.4 | 71.0

11. Secondary Outcome: Percentage of Participants Who Withdrew Because of Lack of Therapeutic Response at Week 97
Description: as for outcome 7
Time Frame: Week 97
Population: ITT Population included all participants who completed double blind period and were re-randomized at Week 24 and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 521 | 372 | 48 | 186
percentage of participants | 1.7 | 3.0 | 4.2 | 1.6

12. Secondary Outcome: Area Under the Serum Concentration Curve of Tocilizumab After First SC Injection or IV Infusion
Time Frame: Week 0: at 6 hours (hr), 24 hr, 48 hr, 96 hr, 120 hr and 168 hr after first dose
Population: Pharmacokinetic-Evaluable Population included all participants who provided at least one evaluable PK sample were included in the pharmacokinetic analysis (PK) analysis. Here, number of participants analyzed who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 17 | 16
microgram*hour/milliliter (mcg*hr/mL) | 1444 (839) | 30988 (9114)

13. Secondary Outcome: Area Under the Serum Concentration Curve of Tocilizumab at Steady State for SC and IV Treatment
Time Frame: Week 20: at 6 hours (hr), 24 hr, 48 hr, 96 hr, 120 hr and 168 hr after dose.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 13 | 13
μg*hr/mL | 7542 (3989) | 41304 (15104)

14. Secondary Outcome: Minimum Serum Concentration (Cmin) of Tocilizumab
Time Frame: Week 0, Week 20: at 6 hours (hr), 24 hr, 48 hr, 96 hr, 120 hr and 168 hr after dose
Population: Pharmacokinetic-Evaluable Population included all participants who provided at least one evaluable PK sample were included in the PK analysis. Here, number of participants analyzed who were evaluable for this outcome measure and 'n' indicates number of participants who were evaluated at specified time point.
Measure: Mean (Standard Deviation); unit: micrgram/milliliter (mcg/mL)
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 17 | 16
micrgram/milliliter (mcg/mL)
  Week 0 (after first dose) (n=17, 16) | 7.48 (4.91) | 6.65 (6.05)
  Week 20 (n=13, 13) | 35.7 (16.2) | 16.0 (10.3)

15. Secondary Outcome: Maximum Serum Concentration (Cmax) of Tocilizumab
Time Frame: Week 0, Week 20: at 6 hours (hr), 24 hr, 48 hr, 96 hr, 120 hr and 168 hr after dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 17 | 16
mcg/mL
  Week 0 (after first dose) (n=17, 16) | 14.7 (8.74) | 180 (40.1)
  Week 20 (n=13, 13) | 52.7 (27.3) | 233 (117)

16. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Tocilizumab
Time Frame: Week 0, Week 20: at 6 hours (hr), 24 hr, 48 hr, 96 hr, 120 hr and 168 hr after dose
Population: as for outcome 14
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Tocilizumab SC | Tocilizumab IV
Number analyzed (Participants) | 17 | 16
hour (hr)
  Week 0 (after first dose) (n=17, 16) | 74 [24 to 121] | 6 [3 to 7]
  Week 20 (n=13, 13) | 70 [0 to 122] | 6 [4 to 46]

17. Secondary Outcome: Change From Baseline in Serum Interleukin-6 (IL-6) Concentration at Week 25
Time Frame: Baseline, Week 25
Population: The ITT-PK population includes all participants who were eligible for the ITT population and provided at least 1 evaluable PK sample in the double blind or open label periods. Here, number of participants analyzed who were evaluable for this outcome measure and 'n' indicates number of participants who were evaluated at specified time point.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 493 | 359 | 46 | 186
picogram/milliliter (pg/mL)
  Baseline (n=493, 359, 46, 186) | 39.04 (55.456) | 52.48 (240.964) | 62.18 (125.081) | 50.07 (161.045)
  Change at Week 25 (n=385, 280, 33, 149) | 34.42 (110.842) | 52.61 (507.157) | 37.54 (93.464) | 44.12 (136.955)

18. Secondary Outcome: Change From Baseline in Serum Soluble Interleukin-6 Receptor (sIL-6R) Concentration at Week 97
Time Frame: Baseline, Week 97
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 504 | 366 | 46 | 186
nanogram/milliliter (ng/mL)
  Baseline (n=504, 366, 46, 186) | 44.53 (35.470) | 45.72 (40.219) | 44.71 (13.068) | 43.28 (16.197)
  Change at Week 97 (n=416, 296, 37,157) | 601.52 (222.141) | 575.75 (244.398) | 569.60 (213.588) | 586.50 (226.915)

19. Secondary Outcome: Percentage of Participants Who Developed Antibodies To Tocilizumab at Week 97
Time Frame: Week 97
Population: The safety population includes all participants who received at least one dose of study drug, whether re-randomized or not, and who had at least one post-dose safety assessment. Here, 'n' indicates number of subjects in the safety population tested by screening assay at any time point.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Number analyzed (Participants) | 629 | 629 | 46 | 184
percentage of participants | 1.3 | 1.0 | 0.0 | 0.5

ADVERSE EVENTS:
Time Frame: Baseline to up to 3 months after last dose of study drug (approximately up to 2 years)
Description: The safety population includes all participants who received at least one dose of study drug, whether re-randomized or not, and who had at least one post-dose safety assessment. Data are included from double blind and open label (OL) periods in the SC and IV arms but only from the OL period in IV-SC and SC-IV switch arms.
Groups:
- Tocilizumab SC Then Tocilizumab IV: Participants who received tocilizumab 162 mg subcutaneous (SC) injection weekly plus placebo to tocilizumab intravenous (IV) infusion every 4 weeks for 24 weeks in double blind treatment period switched to tocilizumab 8 mg/kg IV infusion every 4 weeks for a total of 72 weeks in open label extension period.
  Non-biologic disease-modifying anti-rheumatic drugs (DMARDs) at a stable dose continued throughout the study.
Arm/Group | Tocilizumab SC | Tocilizumab IV | Tocilizumab SC Then Tocilizumab IV | Tocilizumab IV Then Tocilizumab SC
Serious Adverse Events (participants affected / at risk) | 88/631 | 80/631 | 6/48 | 21/186
Other Adverse Events (participants affected / at risk) | 488/631 | 430/631 | 29/48 | 118/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab SC (N=631) | Tocilizumab IV (N=631) | Tocilizumab SC Then Tocilizumab IV (N=48) | Tocilizumab IV Then Tocilizumab SC (N=186)
Pneumonia (Infections and infestations) | 4 | 6 | 0 | 4
Cellulitis (Infections and infestations) | 8 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 0 | 0
Septic Shock (Infections and infestations) | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 3 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 2 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bone tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Burkholderia pseudomallei infection (Infections and infestations) | 0 | 0 | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Pericolic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Whipple's disease (Infections and infestations) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 3 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 0 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Adrenal gland injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Sphincter of oddi dysfunction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 1 | 0 | 0
Amyloidosis (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Device dislocation (General disorders) | 1 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Ischaemic ulcer (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 0
Amaurosis (Eye disorders) | 1 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab SC (N=631) | Tocilizumab IV (N=631) | Tocilizumab SC Then Tocilizumab IV (N=48) | Tocilizumab IV Then Tocilizumab SC (N=186)
Upper respiratory tract infection (Infections and infestations) | 122 | 130 | 8 | 33
Nasopharyngitis (Infections and infestations) | 88 | 68 | 7 | 26
Urinary tract infection (Infections and infestations) | 67 | 53 | 4 | 15
Alanine aminotransferase increased (Investigations) | 188 | 140 | 7 | 29
Aspartate aminotransferase increased (Investigations) | 135 | 96 | 3 | 14
Hypertension (Vascular disorders) | 49 | 65 | 4 | 8
Headache (Nervous system disorders) | 46 | 41 | 3 | 9
Bronchitis (Infections and infestations) | 44 | 35 | 2 | 6
Gastroenteritis (Infections and infestations) | 41 | 26 | 3 | 6
Pharyngitis (Infections and infestations) | 23 | 39 | 2 | 4
Sinusitis (Infections and infestations) | 33 | 19 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 34 | 2 | 9
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 29 | 26 | 3 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 28 | 3 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 11 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 55 | 39 | 1 | 14
Nausea (Gastrointestinal disorders) | 35 | 40 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 62 | 50 | 2 | 13
Fall (Injury, poisoning and procedural complications) | 33 | 25 | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 32 | 27 | 1 | 2
Injection site erythema (General disorders) | 33 | 5 | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.